CLINICAL TRIAL: NCT01999920
Title: Vilazodone for Separation Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #6856
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Separation Anxiety Disorder
Keywords: Adult separation anxiety disorder; ASAD
MeSH Terms: conditions — Anxiety, Separation | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vilazodone (Experimental): Vilazodone treatment. Dosage will begin at 10mg/day and will be increased to 20mg/day after 1 week, and 40mg/day after two weeks (optional). Dosage can be held steady or lowered at any time during the study as clinically indicated in the event of adverse effects. Twelve weeks of treatment, total.
  Interventions: Drug: Vilazodone
- Placebo (Placebo Comparator): Pill placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vilazodone — 10mg to 40mg per day for 12 weeks
  Other Names: Viibryd (brand name)
  Arms: Vilazodone
Drug: Placebo — One to two pills per day for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Vilazodone (Viibryd), an SSRI and 5HT1a receptor agonist, is effective in treating Adult Separation Anxiety Disorder over a 12-week treatment course.

DETAILED DESCRIPTION:
In this randomized clinical trial, 40 adults with a principal diagnosis of Adult Separation Anxiety Disorder (ASAD) and no major depression or substance abuse disorders will be randomized to 12 weeks of treatment with vilazodone (flexibly dosed) or matched pill placebo. Outcome will be assessed in respect to symptomatic improvement, quality of life, adverse events and safety.

ELIGIBILITY:
Inclusion Criteria:

* Current primary (most clinically significant) diagnosis of DSM5 ASAD
* Able to give consent, fluent in English

Exclusion Criteria:

* Past or current DSM-IV diagnosis of any psychotic disorder; organic mental disorder or other cognitive disorder; bipolar disorder; or antisocial personality disorder. Current MDD of moderate or greater severity. Any other current primary Axis I disorder.
* Recent history (past 3 months) of substance or alcohol abuse or dependence (other than nicotine or caffeine)
* Suicidal ideation or behavior (in the past year) that poses a significant danger to the subject
* Medical illness that could significantly increase risk of vilazodone treatment or interfere with assessment of diagnosis or treatment response, including organic brain impairment from stroke, CNS tumor, or demyelinating disease; renal impairment; diabetes mellitus
* Current or past history of seizure disorder (except febrile seizure in childhood)
* History of non-response to ≥ 2 serotonergic reuptake inhibitor antidepressants (SSRIs and/or SNRIs) for the treatment of ASAD after adequate treatment trials (adequate treatment is defined as at least 8 weeks at an adequate dose[s] based on approved package insert recommendations)
* Currently taking medication which has been effective for patient's ASAD
* For patients taking any ineffective psychoactive drug or herbal remedy, inability to tolerate or unwillingness to accept a drug-free period prior to beginning the study of 2 weeks or 5 half-lives (whichever is longer) before beginning study treatment, or ever having been treated with a depot antipsychotic. Fluoxetine washout period will be at least 5 weeks.
* Requiring concomitant treatment with any prohibited medications, supplements, or herbal remedies, except for zolpidem, or zolpidem extended release for insomnia, which may be continued provided the medication has been used in a consistent manner for 4 weeks prior to randomization
* History of intolerance or hypersensitivity to vilazodone, SNRIs or SSRIs
* History of light therapy, electroconvulsive therapy, vagus nerve stimulation, transcranial magnetic stimulation, or any other experimental procedure for central nervous system disorders within 6 months of beginning this study
* Pregnancy, lactation; for women of childbearing potential, not using an effective birth control method (e.g., oral contraceptive or double barrier method) for the duration of the study
* Current formal psychotherapy initiated within 3 months of beginning this study. This includes: psychodynamic, cognitive-behavioral and interpersonal therapies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shear K, Jin R, Ruscio AM, Walters EE, Kessler RC. Prevalence and correlates of estimated DSM-IV child and adult separation anxiety disorder in the National Comorbidity Survey Replication. Am J Psychiatry. 2006 Jun;163(6):1074-83. doi: 10.1176/ajp.2006.163.6.1074. PMID 16741209
- [Background] Winslow JT, Insel TR. Serotonergic modulation of the rat pup ultrasonic isolation call: studies with 5HT1 and 5HT2 subtype-selective agonists and antagonists. Psychopharmacology (Berl). 1991;105(4):513-20. doi: 10.1007/BF02244372. PMID 1771219
- [Background] Simpson BS, Landsberg GM, Reisner IR, Ciribassi JJ, Horwitz D, Houpt KA, Kroll TL, Luescher A, Moffat KS, Douglass G, Robertson-Plouch C, Veenhuizen MF, Zimmerman A, Clark TP. Effects of reconcile (fluoxetine) chewable tablets plus behavior management for canine separation anxiety. Vet Ther. 2007 Spring;8(1):18-31. PMID 17447222
- [Background] Walkup JT, Albano AM, Piacentini J, Birmaher B, Compton SN, Sherrill JT, Ginsburg GS, Rynn MA, McCracken J, Waslick B, Iyengar S, March JS, Kendall PC. Cognitive behavioral therapy, sertraline, or a combination in childhood anxiety. N Engl J Med. 2008 Dec 25;359(26):2753-66. doi: 10.1056/NEJMoa0804633. Epub 2008 Oct 30. PMID 18974308
- [Background] Fluvoxamine for the treatment of anxiety disorders in children and adolescents. The Research Unit on Pediatric Psychopharmacology Anxiety Study Group. N Engl J Med. 2001 Apr 26;344(17):1279-85. doi: 10.1056/NEJM200104263441703. PMID 11323729
- [Derived] Schneier FR, Moskow DM, Choo TH, Galfalvy H, Campeas R, Sanchez-Lacay A. A randomized controlled pilot trial of vilazodone for adult separation anxiety disorder. Depress Anxiety. 2017 Dec;34(12):1085-1095. doi: 10.1002/da.22693. Epub 2017 Oct 25. PMID 29071764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vilazodone | Placebo
Started | 13 | 11
Completed | 7 | 9
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Population: Subjects with adult separation anxiety disorder
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilazodone | Placebo | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (14.2) | 32.9 (15.6) | 35.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 9 | 3 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Hamilton Depression Rating Scale 17-item [Mean (Standard Deviation); unit: units on a scale] — (10 min) Hamilton Rating Scale for Depression (Hamilton, 1960) This standard scale will be used to assess severity of depression, from 0 (least depression) to 50 (greatest depression
  units on a scale | 11.5 (6.3) | 9.3 (5.0) | 10.5 (5.7)
Attachment Style Questionnaire [Mean (Standard Deviation); unit: units on a scale] — (15 min) Attachment Style Questionnaire (Feeney at al., 1994) 40 items relating to quality of adult relationships. Questionnaire includes questions concerning Confidence (8 items, minimum score=8, maximum score=48), Discomfort (10 items, minimum score=10, maximum score=60), Relationships as Secondary (7 items, minimum score=7, maximum score=42), Need for Approval (7 items, minimum score=7, maximum score =42), and Preoccupation with Relationships (8 items, minimum score = 8, maximum score=48), each self-rated on a six-point scale, each self-rated from 1 (totally disagree) to 6 (totally agree)
  units on a scale
    Confidence | 30.5 (5.3) | 25.3 (9.3) | 28.1 (7.7)
    Discomfort with Closeness | 38.2 (8.9) | 46.9 (7.7) | 42.2 (9.3)
    Relationships as Secondary | 17.4 (6.0) | 19.0 (5.9) | 18.1 (5.9)
    Need for Approval | 23.8 (4.6) | 26.1 (8.8) | 24.8 (6.8)
    Preoccupation with Relationships | 34.4 (5.1) | 33.6 (6.3) | 34.0 (5.6)
Quality of Life Enjoyment & Satisfaction Questionnaire [Mean (Standard Deviation); unit: units on a scale] — (10 min) Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q, Endicott et al, 1993): self-rated assessment of quality of life. 16 items related to life quality, each rated on a score of 1 (very poor) to 5 (very good), with a minimum total score of 16, and a maximum total score of 80.
  units on a scale | 46.5 (12.1) | 55.4 (22.2) | 50.6 (17.7)
Structured Clinical Interview for Separation Anxiety Disorder [Mean (Standard Deviation); unit: units on a scale] — Structured Clinical Interview for Separation Anxiety Disorder modified for DSM-5. The eight separation anxiety disorder criteria are each rated on a 0-2 scale for past week time frame. Scores on each of the eight items are summed to produce a total score (range 0 - 16). A higher total score indicates higher symptoms of separation anxiety.
  units on a scale | 10.8 (2.6) | 10.2 (2.5) | 10.5 (2.5)
Adult Separation Anxiety - 27 Scale [Mean (Standard Deviation); unit: units on a scale] — (15 min) Adult Separation Anxiety - 27 Scale 27 items pertaining to adult separation anxiety, each self-rated on a four-point scale, 0=best, 3=worse. Minimum Total Score=0 (better); Maximum Total Score = 81 (worse)
  units on a scale | 44.3 (15.1) | 52.0 (13.6) | 47.8 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Improvement Scale
Description: Clinical Global Impression-Improvement Scale rating at week 12 A quickly administered and widely used observer rating, with ratings from 1 (very much improved) to 7 (very much worse). "Responder" is a score of 1 or 2.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 13 | 11
Participants | 7 | 4
Statistical Analysis 1: Comparison: Vilazodone vs Placebo; Test type: Superiority; p = .064, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline Hamilton Rating Scale for Depression 17-item Total Score
Description: This standard scale will be used to assess severity of depression, looking at change in total score from baseline to week 12, rating severity of depression on a scale from 0 (least depression) to 50 (greatest depression).
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 13 | 11
units on a scale | 3.7 (3.2) | 8.4 (7.2)
Statistical Analysis 1: Comparison: Vilazodone vs Placebo; Test type: Superiority; p = 0.11, Mixed Models Analysis; Standard error = 5.50, 95% CI 2-sided [-1.32 to 12.32], Standard Error of Mean 3.13

3. Secondary Outcome: Change From Baseline in Attachment Style Questionnaire Score
Description: Measure Description: (15 min) Attachment Style Questionnaire (Feeney at al., 1994) 40 items relating to quality of adult relationships. Questionnaire includes questions concerning Confidence (8 items, minimum score=8, maximum score=48), Discomfort (10 items, minimum score=10, maximum score=60), Relationships as Secondary (7 items, minimum score=7, maximum score=42), Need for Approval (7 items, minimum score=7, maximum score =42), and Preoccupation with Relationships (8 items, minimum score = 8, maximum score=48), each self-rated on a six-point scale, each self-rated from 1 (totally disagree) to 6 (totally agree).
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 13 | 11
units on a scale
  Confidence | 32.3 (7.3) | 26.9 (10.3)
  Discomfort with Closeness | 35.6 (5.9) | 42.3 (6.9)
  Relationships as Secondary | 16.3 (4.3) | 20.7 (9.1)
  Need for Approval | 20.6 (3.2) | 23.6 (8.0)
  Preoccupation with Relationships | 30.0 (6.0) | 32.1 (7.8)
Statistical Analysis 1: Comparison: Vilazodone vs Placebo; Confidence variable; Test type: Superiority; p = 0.89, Mixed Models Analysis; Standard error = 0.34, 95% CI 2-sided [-4.85 to 5.53], Standard Error of Mean 2.44
Statistical Analysis 2: Comparison: Vilazodone vs Placebo; Discomfort with Closeness variable; Test type: Superiority; p = 0.79, Mixed Models Analysis; Standard error = 1.18, 95% CI 2-sided [-8.21 to 10.58], Standard Error of Mean 4.41
Statistical Analysis 3: Comparison: Vilazodone vs Placebo; Relationships as Secondary variable; Test type: Superiority; p = 0.31, Mixed Models Analysis; Standard error = 3.94, 95% CI 2-sided [-4.12 to 12.01], Standard Error of Mean 3.79
Statistical Analysis 4: Comparison: Vilazodone vs Placebo; Need for Approval variable; Test type: Superiority; p = 0.10, Mixed Models Analysis; Standard error = -2.60, 95% CI 2-sided [-5.79 to 0.58], Standard Error of Mean 1.49
Statistical Analysis 5: Comparison: Vilazodone vs Placebo; Preoccupation with Relationships variable; Test type: Superiority; p = 0.80, Mixed Models Analysis; Standard error = 0.71, 95% CI 2-sided [-5.30 to 6.72], Standard Error of Mean 2.82

4. Secondary Outcome: Change From Baseline in Quality of Life Enjoyment & Satisfaction Questionnaire
Description: Measure Description: (10 min) Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q, Endicott et al, 1993): self-rated assessment of quality of life. 16 items related to life quality, each rated on a score of 1 (very poor) to 5 (very good), with a minimum total score of 16, and a maximum total score of 80.
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 13 | 11
units on a scale | 68.9 (9.8) | 47.8 (31.0)
Statistical Analysis 1: Comparison: Vilazodone vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis; Standard error = -19.91, 95% CI 2-sided [-34.23 to -5.58], Standard Error of Mean 6.99

5. Secondary Outcome: Change From Baseline on Structured Clinical Interview for Separation Anxiety Disorder
Description: The Structured Clinical Interview for Separation Anxiety Disorder was modified for DSM-5. The eight separation anxiety disorder criteria are rated for both childhood (rated at baseline only) and past week time frames, scored as 0 (not at all), 1 (sometimes), 2 (often) or ? (don't recall). In keeping with the DSM-5 guidelines, endorsement of three or more of the eight criterion symptoms (symptoms rated as '2' or 'often') is used as a threshold to determine categorical (yes/no) diagnosis of separation anxiety disorder. Scores on each of the eight items are also summed to produce a continuous measure of separation anxiety symptoms experienced during childhood and adulthood (range for each scale=0-16).
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 13 | 11
units on a scale | 3.1 (2.4) | 5.0 (3.5)
Statistical Analysis 1: Comparison: Vilazodone vs Placebo; Test type: Superiority; p = 0.026, Mixed Models Analysis; Standard error = 3.29, 95% CI 2-sided [0.42 to 6.16], Standard Error of Mean 1.43

6. Secondary Outcome: Change From Baseline on Adult Separation Anxiety - 27 Scale
Description: Measure Description: (15 min) Adult Separation Anxiety - 27 Scale 27 items pertaining to adult separation anxiety, each self-rated on a four-point scale, 0=best, 3=worse. Minimum Total Score=0 (better); Maximum Total Score = 81 (worse)
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 13 | 11
units on a scale | 14.4 (12.6) | 40.6 (19.2)
Statistical Analysis 1: Comparison: Vilazodone vs Placebo; Test type: Superiority; p = 0.01, Mixed Models Analysis; Standard error = 21.38, 95% CI 2-sided [5.64 to 37.11], Standard Error of Mean 7.65

ADVERSE EVENTS:
Time Frame: Baseline to week 12
Arm/Group | Vilazodone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 13/13 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vilazodone (N=13) | Placebo (N=11)
Headache (Nervous system disorders) | 6 | 3
Heartburn (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2
Decreased Appetite (Gastrointestinal disorders) | 4 | 2
Increased Appetite (Gastrointestinal disorders) | 6 | 5
Dry Mouth (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea/Gas (Gastrointestinal disorders) | 4 | 2
Excessive Sweating (Skin and subcutaneous tissue disorders) | 2 | 2
Skin Problems (Skin and subcutaneous tissue disorders) | 1 | 2
Bruising Easily (Blood and lymphatic system disorders) | 0 | 3
Restlessness (Nervous system disorders) | 3 | 3
Tremor (Nervous system disorders) | 1 | 3
Impaired Coordination (Nervous system disorders) | 1 | 3
Insomnia (General disorders) | 5 | 3
Fatigue (General disorders) | 3 | 5
Somnolence (Nervous system disorders) | 2 | 6
Decreased Libido (men) (Reproductive system and breast disorders) | 2 | 0
Decreased Libido (women) (Reproductive system and breast disorders) | 1 | 4
Sexual Dysfunction (men) (Reproductive system and breast disorders) | 2 | 0
Sexual Dysfunction (women) (Reproductive system and breast disorders) | 4 | 4
Blurry Vision (Eye disorders) | 1 | 5
Lightheadedness (Nervous system disorders) | 6 | 6
Forgetfulness (Nervous system disorders) | 1 | 2
Impaired Concentration (Nervous system disorders) | 5 | 5
Apathy (Nervous system disorders) | 3 | 3
Nervousness (Nervous system disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT01999920/SAP_000.pdf
  • Informed Consent Form (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT01999920/ICF_001.pdf
  • Study Protocol (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT01999920/Prot_002.pdf